CLINICAL TRIAL: NCT01808105
Title: Growth and Tolerance of Young Infants Fed Infant Formulas
Brief Title: Growth and Tolerance of Infants Fed Infant Formulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: AL06
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Growth and Tolerance
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Human Milk (Other): Reference group, breast feeding ad libitum
  Interventions: Other: Human Milk
- Control Formula (Active Comparator): Ready to feed infant formula, feed ad libitum
  Interventions: Other: Control Formula
- Experimental Formula 1 (Experimental): Ready to feed infant formula with human milk oligosaccharides, feed ad libitum
  Interventions: Other: Experimental Formula 1
- Experimental Formula 2 (Experimental): Ready to feed infant formula with human milk oligosaccharides, feed ad libitum
  Interventions: Other: Experimental Formula 2

INTERVENTIONS:
Other: Control Formula — Feeding ad libitum
  Other Names: Commercially available Infant Formula
  Arms: Control Formula
Other: Experimental Formula 1 — Feeding ad libitum
  Arms: Experimental Formula 1
Other: Experimental Formula 2 — Feeding ad libitum
  Arms: Experimental Formula 2
Other: Human Milk — Feeding ad libitum
  Other Names: Breast feeding group
  Arms: Human Milk

SUMMARY:
To evaluate growth and tolerance of healthy term infants fed experimental infant formulas, a commercial infant formula and human breast milk.

ELIGIBILITY:
Inclusion Criteria:

* Singleton from full term birth with a gestational age 37-42 weeks
* Birth weight > 2490 g (~5 lbs 8 oz)
* Between 0 and 5 days of age
* Smoke-free home (no smoking in the house dwelling), and mothers in the breast-fed group are prohibited from smoking during the study period
* Parent(s) of formula-fed infants have elected not to breastfeed and confirm that their infant has been exclusively formula-fed since birth and confirm their intention is to exclusively feed their infant study infant formula for the duration of the study,
* Parent(s) of human milk-fed infants have elected to breastfeed and confirm that their infant has been exclusively human milk-fed (not donor milk) since birth and confirm their intention is to continue to exclusively feed human milk with vitamin/mineral supplementation for the duration of the study
* No administration vitamin or mineral supplements (excluding vitamin or mineral supplements containing vitamin D, if recommended by a healthcare professional), solid foods or juices to infants from enrollment through the duration of the study, unless instructed otherwise by their healthcare professional

Exclusion Criteria:

* Adverse maternal, fetal or infant medical history that has potential effects on tolerance, growth, and/or development
* Infants using medications, home remedies, herbal preparations, probiotics or rehydration fluids that might affect gastrointestinal (GI) tolerance may not be enrolled
* Treatment with antibiotics
* Mother intends to use a combination of breast and formula feeding

Max Age: 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 424 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Weight | Study Day (SD) 14 - 119
  Weight gain per day

SECONDARY OUTCOMES:
Stool Characteristics | Study Day (SD) 1-28; 3 Day Records prior to SD 42, 84 and 119 visits
  Stool consistency and number per day
Feeding Tolerance | Study Day (SD) 1-28; 3 Day Records prior to SD 42, 84 and 119 visits
  % of feedings with spit up associated with feeding
Length | Study Day (SD) 1, 14, 28, 42, 84 and 119 visits
  Length and interval length gain per day
Head Circumference | Study Day (SD) 1, 14, 28, 42, 84 and 119 visits
  Head circumference (HC) and interval HC gain per day

OTHER OUTCOMES:
Study Formula Intake | Study Day (SD) 1-28; 3 Day Records prior to SD 42, 84 and 119 visits
  Average volume of study formula intake and average number of study formula feedings per day
Oligosaccharides | Study Day (SD) 42 and 119 visits
  Infant urine sample

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Williams, MPH, Study Chair — Abbott Nutrition
Locations (25):
- United States (23):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Alabama Clinical Therapeutics, Dothan, Alabama
  - W.O.M.B Watching Over Mothers and Babies, Tucson, Arizona
  - Clinical Research Advantage/Colorado Springs Health Partners, Colorado Springs, Colorado
  - Norwich Pediatric Group, PC, Norwich, Connecticut
  - Atlantic Clinical Research Collaborative, Boynton Beach, Florida
  - Lake Mary Pediatrics, Orange City, Florida
  - SCORE Physician Alliance, LLC, St. Petersburg, Florida
  - USF, College of Medicine, Dept of Pediatrics, Tampa, Florida
  - Southeast Regional Research Group (SERRG), Columbus, Georgia
  - PediaResearch, LLC, Evansville, Indiana
  - Northpoint Pediatrics, LLC, Indianapolis, Indiana
  - Lafayette Clinical Research, Lafayette, Indiana
  - Women's Clinic of Lincoln, PC, Lincoln, Nebraska
  - MetroHealth Medical Center, Cleveland, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - Ohio Pediatric Research Association, Inc, Dayton, Ohio
  - Institute of Clinical Research, Mayfield Heights, Ohio
  - Clinical Trials of America, Eugene, Oregon
  - Red Lion Pediatrics, Philadelphia, Pennsylvania
  - Sanford Research, Sioux Falls, South Dakota
  - Tanner Memorial Clinic, Layton, Utah
  - Rockwood Clinic, PS, Spokane, Washington
- Puerto Rico (2):
  - Clinical Research Puerto Rico, Guayama
  - Ponce School of Medicine/ CAIMED Center, Ponce

REFERENCES:
- [Derived] Hill DR, Buck RH. Infants Fed Breastmilk or 2'-FL Supplemented Formula Have Similar Systemic Levels of Microbiota-Derived Secondary Bile Acids. Nutrients. 2023 May 17;15(10):2339. doi: 10.3390/nu15102339. PMID 37242222
- [Derived] Goehring KC, Marriage BJ, Oliver JS, Wilder JA, Barrett EG, Buck RH. Similar to Those Who Are Breastfed, Infants Fed a Formula Containing 2'-Fucosyllactose Have Lower Inflammatory Cytokines in a Randomized Controlled Trial. J Nutr. 2016 Dec;146(12):2559-2566. doi: 10.3945/jn.116.236919. Epub 2016 Oct 26. PMID 27798337